CLINICAL TRIAL: NCT06404242
Title: Plaque Characteristics From Vessel Wall Magnetic Resonance Imaging Predict Recurrent Stroke in Ischemic Stroke Patients Due to Middle Cerebral Artery Stenosis
Brief Title: Plaque Characteristics Predict Recurrent Stroke in MCA Stroke Patients
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Principal Investigator, Dao Duy Khoa, Principal Investigator, University Medical Center Ho Chi Minh City (UMC)
Other Study IDs: IRB-VN01002
Record Dates: First submitted 2024-04-29; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Stroke, Ischemic; Atherosclerosis, Cerebral
MeSH Terms: conditions — Ischemic Stroke; Intracranial Arteriosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MCA stroke patient: The investigators would include patients who had ischemic stroke due to middle cerebral artery (MCA) stenosis (>50%). The investigators collect plaque characteristics such as plaque enhancement, T1 hyperintense, remodeling ratio, surface irregularity, correlation with the origin of perforating branches, percent stenosis, upstream angle, and downstream angle. The patients were followed up for stroke recurrence for 6 months.
  For each culprit-plaque characteristic, the investigators would divide the patients into groups of patients with culprit-plaque characteristics and groups without culprit-plaque characteristics. The two groups will compare the type of ischemic lesions and the recurrent stroke rate in the same vascular territory. These results will be presented by Kaplan-Meier curve and binary logistic regression.

SUMMARY:
The epidemiology of TOAST classification in Asian patients seems to differ due to the higher rates of large-artery atherosclerosis. The complex pathology of atherosclerosis could lead to recurrent stroke, including shear stress on the endothelium, disturbance of the flow, occlusion at the origin of the perforating artery, and other complications (plaque inflammation, plaque hemorrhage, plaque rupture) that could lead to stroke and recurrent stroke. Therefore, The exact determination of the etiology of stroke due to atherosclerosis is the most critical factor for treatment and prognostic. On the other hand, HR-MRI could be a useful imaging modality to evaluate the characteristics of plaque in stroke patients due to atherosclerosis stenosis, which will help us find out the etiology of stroke. Previous studies have demonstrated its prognosis value in predicting recurrent stroke in the same vascular territory. The investigators hypothesize that with an appropriate evaluation, HR-MRI could help to predict recurrent stroke in the same vascular territory in patients with high-risk plaque characteristics on HR-MRI. These findings could contribute to individual treatment according to etiology.

The investigators intend to conduct a study to determine the correlation between plaque characteristics and recurrent stroke in the same vascular territory in ischemic stroke patients due to middle cerebral artery stenosis.

DETAILED DESCRIPTION:
The epidemiology of TOAST classification in Asian patients seems to differ due to the higher rates of large-artery atherosclerosis 1. The complex pathology of atherosclerosis could lead to recurrent stroke, including shear stress on the endothelium, disturbance of the flow, occlusion at the origin of the perforating artery, and other complications (plaque inflammation, plaque hemorrhage, plaque rupture) that could lead to stroke and recurrent stroke 2. Therefore, The exact determination of the etiology of stroke due to atherosclerosis is the most critical factor for treatment and prognostic. On the other hand, HR-MRI could be a useful imaging modality to evaluate the characteristics of plaque in stroke patients due to atherosclerosis stenosis, which will help us find out the etiology of stroke 3. Previous studies have demonstrated its prognosis value in predicting recurrent stroke in the same vascular territory 4. The investigators hypothesize that with an appropriate evaluation, HR-MRI could help to predict recurrent stroke in the same vascular territory in patients with high-risk plaque characteristics on HR-MRI. These findings could contribute to individual treatment according to etiology 5,6.

The investigators intend to conduct a study to determine the correlation between plaque characteristics and recurrent stroke in the same vascular territory in ischemic stroke patients due to middle cerebral artery stenosis

ELIGIBILITY:
Inclusion Criteria:

* Patients who had a first-time ischemic stroke due to MCA atherosclerosis stenosis more than 50% and admitted to our hospital within 7 days after onset.
* Patients are more than 45 years old.
* Patients had HR-MRI and have done the full stroke workup (including carotid duplex scanning, fasting lipid profile, Holter ECG 24 hours, cardiac ultrasound,...)

Exclusion Criteria:

* Patients also have stenosis of the carotid artery (more than 50%) on the same side of ischemic stroke.
* Patients also have an ischemic stroke in territories other than MCA territory.
* Patients had any characteristics that suggested other causes for their stenosis, including moyamoya, dissection, and inflammation on their MRI and HR-MRI.
* Patients with evidence suggestive of cardioembolism (Atrial fibrillation, decreased EF <50%, recent heart attack in 3 weeks, rheumatic valvular heart disease, dilated cardiopathy, sick sinus syndrome, infective endocarditis).
* Any signs suggestive of autoimmune disease or increased coagulation state.
* Patients with severe concomitant disease could affect the 6-month follow-up of the patients.

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators would include patients who had ischemic stroke due to middle cerebral artery (MCA) stenosis (>50%)
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The rate of recurrent stroke at the same vascular territory for each culprit-plaque characteristic on HR-MRI | 04/2024-02/2026
  The investigators will determine the rate of recurrent stroke based on the clinical presentation in combination with the MRI lesion if the patient has symptoms suggestive of recurrent stroke.

SECONDARY OUTCOMES:
Determine the rate of plaque characteristics | 04/2024-02/2026
  The investigators will examine the plaque characteristics of high-resolution MRI, including plaque enhancement, T1 hyperintense, remodeling ratio, surface irregularity, correlation with the origin of perforating branches, upstream angle, and downstream angle
Determine the correlation between plaque characteristics and type of ischemic lesions (stroke mechanism) for each of culprit-plaque characteristics on MRI | 04/2024-02/2026
  The investigators will divide the type of ischemic stroke into Artery-to-Artery Embolic Infarction or non Artery-to-Artery Embolic Infarction (including Occlusion of perforating branches, hypoperfusion, or combination).

CONTACTS AND LOCATIONS:
Overall Officials: Khoa Dao, MD, Principal Investigator — University Medical Center Ho Chi Minh City
Locations (1):
- University Medical Center Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
When there is an appropriate request, the investigators will consider and provide anonymous data
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be available after the study has finished for at least 1 year and will be available for 3 years
Access Criteria: Upon reasonable request

REFERENCES:
- [Background] Bang OY. Considerations When Subtyping Ischemic Stroke in Asian Patients. J Clin Neurol. 2016 Apr;12(2):129-36. doi: 10.3988/jcn.2016.12.2.129. Epub 2016 Jan 28. PMID 26833987
- [Background] Wong KS, Caplan LR, Kim JS. Stroke Mechanisms. Front Neurol Neurosci. 2016;40:58-71. doi: 10.1159/000448302. Epub 2016 Dec 2. PMID 27960181
- [Background] Song JW, Pavlou A, Xiao J, Kasner SE, Fan Z, Messe SR. Vessel Wall Magnetic Resonance Imaging Biomarkers of Symptomatic Intracranial Atherosclerosis: A Meta-Analysis. Stroke. 2021 Jan;52(1):193-202. doi: 10.1161/STROKEAHA.120.031480. Epub 2020 Dec 2. PMID 33370193
- [Background] Wu F, Song H, Ma Q, Xiao J, Jiang T, Huang X, Bi X, Guo X, Li D, Yang Q, Ji X, Fan Z; WISP Investigators. Hyperintense Plaque on Intracranial Vessel Wall Magnetic Resonance Imaging as a Predictor of Artery-to-Artery Embolic Infarction. Stroke. 2018 Apr;49(4):905-911. doi: 10.1161/STROKEAHA.117.020046. Epub 2018 Mar 14. PMID 29540606
- [Background] Johnston SC, Easton JD, Farrant M, Barsan W, Conwit RA, Elm JJ, Kim AS, Lindblad AS, Palesch YY; Clinical Research Collaboration, Neurological Emergencies Treatment Trials Network, and the POINT Investigators. Clopidogrel and Aspirin in Acute Ischemic Stroke and High-Risk TIA. N Engl J Med. 2018 Jul 19;379(3):215-225. doi: 10.1056/NEJMoa1800410. Epub 2018 May 16. PMID 29766750
- [Background] Wang Y, Wang Y, Zhao X, Liu L, Wang D, Wang C, Wang C, Li H, Meng X, Cui L, Jia J, Dong Q, Xu A, Zeng J, Li Y, Wang Z, Xia H, Johnston SC; CHANCE Investigators. Clopidogrel with aspirin in acute minor stroke or transient ischemic attack. N Engl J Med. 2013 Jul 4;369(1):11-9. doi: 10.1056/NEJMoa1215340. Epub 2013 Jun 26. PMID 23803136
- [Background] Kim JM, Jung KH, Sohn CH, Moon J, Shin JH, Park J, Lee SH, Han MH, Roh JK. Intracranial plaque enhancement from high resolution vessel wall magnetic resonance imaging predicts stroke recurrence. Int J Stroke. 2016 Feb;11(2):171-9. doi: 10.1177/1747493015609775. PMID 26783308
- [Background] Leung TW, Wang L, Zou X, Soo Y, Pu Y, Ip HL, Chan A, Au LWC, Fan F, Ma SH, Ip B, Ma K, Lau AY, Leung H, Hui KF, Li R, Li SH, Fu M, Fong WC, Liu J, Mok V, Wong KSL, Miao Z, Ma N, Yu SCH, Leng X. Plaque morphology in acute symptomatic intracranial atherosclerotic disease. J Neurol Neurosurg Psychiatry. 2020 Nov 25;92(4):370-6. doi: 10.1136/jnnp-2020-325027. Online ahead of print. PMID 33239439